CLINICAL TRIAL: NCT05929690
Title: A Feasibility Trial of Self-Acupuncture for Chemotherapy Cancer Patients (SACC Trial)
Brief Title: Feasibility Trial Self-Acupuncture for Chemotherapy Cancer Patients
Acronym: SACC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University College London Hospitals (Other)
Responsible Party: Principal Investigator, John Hughes, Associate Professor, University College London Hospitals
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 152103
Record Dates: First submitted 2023-05-06; First posted 2023-07-03 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Cancer
Keywords: cancer; acupuncture; feasibility trial
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard care plus self-acupuncture (Experimental): Participants randomised to the self-acupuncture arm will be asked to attend a group workshop. All participants will be taught to safely apply acupuncture bilaterally using traditional acupuncture needles to the acupuncture point Stomach 36. If deemed to be clinically appropriate by the acupuncturists, and if patients are willing and able, they will also be taught how to safely needle the acupuncture points Spleen 6 and/or Liver 3 (maximum of six points in total). Participants will be asked to needle the points 2-3 times a week throughout their cancer treatment and for 3 months post treatment.
  Interventions: Other: Self-acupuncture
- Standard care (No Intervention): Chemotherapy patients allocated to standard care will receive no additional treatments. 'Standard care' for all patients will be consistent with current best practice.

INTERVENTIONS:
Other: Self-acupuncture — Participants be taught to safely apply acupuncture bilaterally using traditional acupuncture needles to the acupuncture point Stomach 36. If deemed to be clinically appropriate by the acupuncturists, and if patients are willing and able, they will also be taught how to safely needle the acupuncture points Spleen 6 and/or Liver 3 (maximum of six points in total).
  Arms: Standard care plus self-acupuncture

SUMMARY:
The proposed study will employ a pragmatic mixed methods randomised parallel-group exploratory design to determine the feasibility of delivering self-acupuncture within an NHS cancer care setting. The trial will explore the feasibility and acceptability of all aspects of a definitive clinical trial of teaching cancer patients to self-administer acupuncture to alleviate symptoms of cancer and the side effects of conventional chemotherapy treatment. In addition the feasibility trial will provide preliminary data on effectiveness to inform the sample size calculation for a controlled clinical trial. Patients will be randomly allocated to receive either: 1) self-acupuncture in addition to standard care or 2) standard care alone. Participants randomised to the self-acupuncture arm will be asked to attend a 1.5 hour group workshop delivered by an experienced practitioners and teachers of self-acupuncture. Participants allocated to standard care will be offered training in self-acupuncture once the trial is complete to address any ongoing side effects from their cancer and its treatment. Patients will be recruited at the initiation of their chemotherapy cancer treatment from UCH Macmillan Cancer Centre. Participants will complete baseline outcome measures and be asked to complete follow up outcomes measures at the end of chemotherapy treatment, and 3 months post chemotherapy treatment. At the end of chemotherapy treatment participants will also be asked to take part in a qualitative telephone interview to explore their views on the design of the study and if allocated to self-acupuncture their views on the intervention. At 3 months post chemotherapy treatment those allocated to self-acupuncture will be invited to participate in a second qualitative interview to explore the long-term practice and effects of self-acupuncture. Qualitative interviews will also be conducted with stakeholders (acupuncturists delivering workshops and UCH Macmillan Cancer Centre staff) to explore their views on the feasibility of teaching cancer patients self-acupuncture.

ELIGIBILITY:
Inclusion Criteria:

* Patients due to receive radical (curative) intravenous chemotherapy (any chemotherapy regime).
* Patients of either gender and older than 16 years old.
* Patients with any cancer diagnosis.
* Patients willing to participate in the study and be randomised to one of the two treatment arms.
* Patients willing to attend the self-acupuncture workshop, and self-administer acupuncture, if assigned to the intervention.

Exclusion Criteria:

* Palliative patients.
* Patients unwilling to participate (for instance due to needle phobia).
* Patients currently receiving acupuncture.
* Patients with a platelet count <20 000mm.
* Patients with a white blood cell count <1000mm.
* Patients with severe clotting dysfunction or who bruise spontaneously.
* Patients unable to complete the questionnaires as judged by the investigators.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-11-16 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
European Organization for Research and Treatment of Cancer-Quality of Life Questionnaire-Core 30 Item (EORTC QLQ-C30) | This scale will measure change at baseline and upon completion of chemotherapy treatment (up to 26 weeks later)
  This is a well-validated quality of life questionnaire focusing on functional assessment. The EORTC QLQ-C30 incorporates nine multi-item scales: five functional scales (physical, role, cognitive, emotional, and social); three symptom scales (fatigue, pain, and nausea and vomiting); and a global health and quality-of-life scale.
Multidimensional Fatigue Inventory (MFI) | This scale will measure change at baseline and upon completion of chemotherapy treatment (up to 26 weeks later)
  The MFI is a well-validated scale measuring general fatigue including the dimensions of physical and mental fatigue, activity, and motivation. The questionnaire comprises 20 items for which the person must specify the extent to which the particular statements relates to them on a five-point scale, ranging from Yes, that is true to No, that is not true.
Memorial Symptom Assessment Scale | This scale will measure change at baseline and upon completion of chemotherapy treatment (up to 26 weeks later)
  This is a multidimensional scale which evaluates 32 physical and psychological symptoms associated with cancer and its treatment.
Visual Analogue Scale of Quality of Life | This scale will measure change at baseline and upon completion of chemotherapy treatment (up to 26 weeks later)
  The Visual Analogue Scale (VAS) is a commonly used outcome measurement to monitor variations in patient reported quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- UCH Macmillan Cancer Centre, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No